CLINICAL TRIAL: NCT02493933
Title: Phytoestrogen, NO Donors, N-acetyl Cysteine Add Therapy to Clomiphene
Brief Title: Phytoestrogen, NO Donors, N-acetyl Cysteine Add Therapy to Clomiphene Citrate to Improve Pregnancy Rate in PCO Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Nawara Mohamed Hashish, Assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43-2015
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Phytoestrogens; Acetylcysteine

ARMS (3):
- Phytoestrogen (Active Comparator): Patients received oral PE 120 mg/ day in the form of dry coated tablets (Klimadynon, Bionorica, Germany) 2 tablets three times daily from day 1 to day 12 as adjuvant to CC in the follicular phase of the cycle.
  Interventions: Drug: Phytoestrogens, Isosorbid mononitrate, N-acetyl cysteine
- Isosorbid mononitrate (Active Comparator): Patients received in addition to CC 20 mg Isosorbid mononitrate (ISMN) tablet (EFFOX, Minapharm Co., Egypt under licence of Shwartz pharma,Germany) applied vaginally from day 1 to day 12 of the cycle.
  Interventions: Drug: Phytoestrogens, Isosorbid mononitrate, N-acetyl cysteine
- N-Acetyl cysteine (Active Comparator): Patients received supplementation to CC with NAC 1200 mg/day orally (N-acetyl cysteine, Sedico, Cairo, ARE) sachets 200 mg each, as two sachets thrice daily from day 1 to day 12 of the cycle.
  Interventions: Drug: Phytoestrogens, Isosorbid mononitrate, N-acetyl cysteine

INTERVENTIONS:
Drug: Phytoestrogens, Isosorbid mononitrate, N-acetyl cysteine

SUMMARY:
To evaluate the effect of oral Phytoestrogen or Isosorbid mononitrate or N-acetyl cysteine as an adjuvant to clomiphene citrate on induction of ovulation and pregnancy outcomes in patients with PCOS. In this three-arm open RCT, 240 PCOS infertile women were randomly divided to 3 groups for induction of ovulation. Group A, [PE group, n= 80] patients received CC 100mg/d plus oral Phytoestrogen120 mg/ day and patients in Group B, [ISMN group, n=80] received CC 100 mg/d plus 20 mg Isosorbid mononitrate and Group C, [NAC group, n=80] patients received CC 100 mg/d plus NAC 1200 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. All patients have PCOS.
2. All patients received CC 100 mg/day for 5 days starting from day 5 with successful ovulation as documented by folliculometry and midluteal serum progesterone with no pregnancy achieved.
3. All patients have patent fallopian tubes by Hysterosalpingography.
4. Their husbands have normal semen analysis according to the modified criteria of WHO.
5. All patients have normal serum prolactin and thyroid profile.
6. Any patient having vaginitis was treated before starting induction.

Exclusion Criteria:

1. Other causes of infertility than anovulation.
2. Diabetes or other endocrinological disorders.
3. Age > 40 years.
4. Smoking.
5. Alcohol use.
6. Presence of ovarian cyst >2cm on the second day of the cycle.
7. Patients who have received gonadotrophins in the preceeding 6 months.
8. Patients who have done unilateral or bilateral ovarian drilling.
9. Allergy to PE, NO donors or NAC

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 6 months